CLINICAL TRIAL: NCT01881087
Title: Spinal Anesthesia With Hyperbaric Levobupivacaine 0.75% for Ambulatory Knee Arthroscopy: A Double Blind, Randomized Clinical Trial Comparing Three Low Doses
Brief Title: Spinal Anesthesia With Hyperbaric Levobupivacaine 0.75% for Ambulatory Knee Arthroscopy
Acronym: levobupi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Principal Investigator, Fredy Ariza, Anesthesiologist, Epidemiologist, Fundacion Clinica Valle del Lili
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LevoBupi-003
Record Dates: First submitted 2013-06-16; First posted 2013-06-19 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-04

CONDITIONS: Disorder of Knee; Anesthesia
Keywords: Knee Arthroscopy; Levobupivacaine; Spinal Anesthesia; Motor Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Levo-7.5 mg (Experimental): Hyperbaric Levobupivacaine 0.75% Spinal Administration by a Whitacre Needle 27G. Dosage: 7.5 mg. Single Dose.
  Interventions: Drug: Hyperbaric Levobupivacaine 0.75%
- Levo-9.37 (Experimental): Hyperbaric Levobupivacaine 0.75% Spinal Administration by a Whitacre Needle 27G. Dosage: 9.37 mg. Single Dose.
  Interventions: Drug: Hyperbaric Levobupivacaine 0.75%
- Levo-11.25 (Active Comparator): Hyperbaric Levobupivacaine 0.75% Spinal Administration by a Whitacre Needle 27G. Dosage: 11.25 mg. Single Dose.
  Interventions: Drug: Hyperbaric Levobupivacaine 0.75%

INTERVENTIONS:
Drug: Hyperbaric Levobupivacaine 0.75% — Each 4 ml of the administred solution contains: Chlorhydrate Levogyre Bupivacaine 30 mg, Glucose 290.8 mg and water for injection c.s.
  Other Names: Bupinest 0.75% Pesado

SUMMARY:
The purpose of this study is to evaluate motor block probability throughout time and clinical profile when using three different doses of HLBP 0.75% (7.5, 9.37 and 11.25 mg) by a unilateral spinal block technique.

DETAILED DESCRIPTION:
Previous IRB approval and informed consent, 180 ASA I-II adults under ambulatory knee arthroscopy will be randomly allocated to receive unilateral spinal anesthesia with 7.5 (group Levo-7.5, n=59), 9.37(group Levo-9.37, n=61) and 11.25 (group Levo-11.25, n=60) mg of HLBP 0.75% using a 27-gauge Whitacre needle at a rate of 0.1 ml/ seg. and lateral decubitus position maintained for 5 min after injection.

An independent observer will evaluate motor (modified Bromage scale) and sensory (transcutaneal electrical stimulation at T10, L1, L3, and S1 dermal segments) levels and presence of adverse events immediately after return to supine, at the end of surgery and each 10 min from admission to PACU until home discharge conditions.

Trans-cutaneal electrical stimulation (TES) will be made with a PNS (Ministim® model MS- IV, Organon, Dublin, Irland) using 50-Hz tetanus stimuli for 5 seg. from 10 to 60 mA 3,4.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-64 y.o. scheduled for knee arthroscopy (therapeutic or diagnostic)

Exclusion Criteria:

* Cardiac or pulmonary disease
* Antiplatelet or anticoagulant drugs use during 7 days before surgery
* History of coagulative disorders
* Bilateral procedures

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredy J Ariza, MD., MSc., Principal Investigator — Fundacion Clinica Valle del Lili; Marisol Badiel, MD., MSc., Study Chair — Unidad de Investigaciones Clínicas, Fundación Valle del Lili
Locations (1):
- Fundación Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: Yes
IPD is available if DB is formally requested to the Clinical Research Center of the Fundación Valle del Lili (Info: +57 3319090 Ext 4124. http://www.institutodeinvestigaciones.org/)

REFERENCES:
- See also: http://apps.elsevier.es/watermark/ctl_servlet?_f=10&pident_articulo=90150010&pident_usuario=0&pcontactid=&pident_revista=341&ty=7&accion=L&origen=reuma%20&web=http://www.revcolanest.com.co&lan=es&fichero=341v38n04a90150010pdf001.pdf — http://www.redalyc.org/articulo.oa?id=195119002005

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levo-7.5 mg | Levo-9.37 | Levo-11.25
Started | 60 | 61 | 62
Completed | 59 | 61 | 60
Not Completed | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levo-7.5 mg | Levo-9.37 | Levo-11.25 | Total
Number analyzed (Participants) | 59 | 61 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (13) | 47 (13) | 44 (12) | 44.3 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 32 | 92
  Male | 27 | 33 | 28 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 61 | 60 | 180
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Colombia | 59 | 61 | 60 | 180
Weight [Mean (Standard Deviation); unit: kilograms] | 74.7 (12.3) | 73.3 (11.4) | 75.7 (13.9) | 74.5 (12.5)
Height [Mean (Standard Deviation); unit: centimeters] | 168 (9) | 167 (6) | 168 (9) | 168 (8)

OUTCOME MEASURES:

1. Primary Outcome: Probability of Motor Block
Description: Likelihood Rate of motor block persistence after a dosis of spinal HLBP 0.75%
Time Frame: 200 minutes
Measure: Number; unit: percentage of motor block
Arm/Group | Levo-7.5 mg | Levo-9.37 | Levo-11.25
Number analyzed (Participants) | 59 | 61 | 60
percentage of motor block | 5 | 20 | 27

2. Secondary Outcome: Failed Spinal Block Rate
Description: Failed Spinal Block Rate for each treatment group
Time Frame: 15 minutes after dose
Measure: Count of Participants; unit: Participants
Arm/Group | Levo-7.5 mg | Levo-9.37 | Levo-11.25
Number analyzed (Participants) | 59 | 61 | 60
Participants | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research
Arm/Group | Levo-7.5 mg | Levo-9.37 | Levo-11.25
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/61 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/61 | 0/60
Other Adverse Events (participants affected / at risk) | 0/59 | 0/61 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No